CLINICAL TRIAL: NCT01836640
Title: Developing Plasma DNA as a Surrogate for Tumor Biopsy to Identify Tumor Genetic Alterations in Patients With Advanced Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Primary goal not achievable
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D13100
Record Dates: First submitted 2013-04-16; First posted 2013-04-22 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2013-03

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There are three major subtypes of breast cancer:

1. Hormone receptor positive (contain cells that express the estrogen receptor or progesterone receptor).
2. Tumors that express the epidermal growth factor receptor gene ( HER-2)
3. Triple negative (cancer cells that lack the hormone receptors and the epidermal growth factor receptor gene HER-2.

While effective therapies exist for most cases of breast cancer at first occurrence, many patients eventually exhibit disease that does not respond to all standard breast therapies, particularly in the metastatic setting.

There are therapies that are used to treat other types of cancers with genetic mutations that are in the process of being evaluated for use in breast cancer. The current techniques used for detecting mutations in the genes of breast cancer patients, which can be treated with drugs specific for the genetic mutations, are invasive and identifying effective diagnostic non-invasive procedures are the next challenge for physicians. This study will compare the ability to detect genetic mutations samples from non-invasive procedures such as a blood draw, to more invasive procedures such as tissue taken from a biopsy sample.

There is also a concern with current techniques used to detect genetic mutations that cells from a single tissue sample may not be representative of the types of cells present in all the tumors in the body and therapies selected using a single tissue sample may not be effective for all of the cancer in the body. This study will use blood drawn from participants prior to any drug therapy and compare the genes from this blood to tissue samples from multiple sites of disease.

The study will also compare the genetic profile of the metastatic tumors to the genetic profile of the original breast cancer to determine if there are any changes in the genetics of the tumor cells.

The participants that have newly diagnosed metastatic disease will provide tissue from their primary site of disease via an image guided biopsy. These participants will also provide tissue from at least 2 other distant metastatic sites (lung, pleural/peritoneal, liver, brain, or skin). Each biopsy procedure will attempt to obtain 2-3 samples for research purposes.

Participants that have locally recurrent disease in the breast will have the tissue from the site of re-occurrence biopsied as well as two distant metastatic sites (lung, pleural/peritoneal, liver, brain, or skin). Participants that have either multi-centric disease or bilateral disease will have all tumors sampled with the intention of providing 2-3 samples/tumor for research purposes. Participants with multi-centric and bilateral disease will also have 2 distant sites of distant disease sampled (lung, pleural/peritoneal, liver, brain, or skin).

Prior to any scheduled biopsy procedures all participants will have a blood draw used to examine the genetics of the tumor cells in the blood. The participants will have 8 tubes of blood drawn for the test and then they will proceed onto the tissue sampling portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* 3.1 Radiographic evidence of new or progressive metastatic breast cancer by CT chest/abdomen/pelvis and bone scan, or by PET scan.
* 3.2 Patient must have ≥3 sites of disease involving ≥2 organ sites appropriate for biopsy. Treating physician, in consultation with interventional radiologist as needed, will select sites for potential biopsy (see section 5.2.2 for guidance on evaluable sites.)Histologic documentation of metastatic invasive breast cancer with metastasis to a distant organ site (lung, liver, pleural/peritoneal, skin [if skin, must be determined by treating physician that it is not skin involvement from breast primary or local regional recurrence], and/or bone) by core needle or excisional biopsy.
* 3.3 The subject must agree to undergo and be able to tolerate the research biopsy(ies) and blood draw.
* 3.4 Prior chemotherapy, endocrine therapy, or radiotherapy with therapeutic intent is allowed in the metastatic setting. However, for patients currently receiving such treatment(s), archived tumor specimens will not count towards the required biopsy of 3 tumors
* 3.5 Women or men > age 18.
* 3.6 Ability to give informed consent.
* 3.7 Normal Prothrombin Time/International Normalized Ratio within 30 days of any diagnostic biopsies, or if patient is on anticoagulation therapy, approval is required by provider doing the biopsy.
* 3.8 Negative pregnancy test or beyond reproductive potential.
* 3.9 Medical evaluation by medical oncology within 4 weeks.
* 3.10 Previous but not current smokers are eligible if they have not smoked for more than 10 years and have less than 25 pk yr smoking history, see exclusion criterion 3.14.

Exclusion Criteria:

3.12 Poor venous access (unable to tolerate large-gauge needle).

3.13 Unable to tolerate blood draw or research biopsy procedures.

3.14 Current smokers or smoked at all within the last 10 years, or have a lifetime smoking history greater than 25 pack-years. (One pack year is equal to smoking 1 pack per day for 1 year; 5 pack years = one pack/day for 5 yrs, or ½ pack/day for 10 yrs, etc.). There is evidence that smoking increases the likelihood of detecting mutations in cancer-related genes in plasma DNA in healthy individuals (i.e., who do not have detectable cancer) (15, 16). We wish to avoid detecting such genetic lesions in this pilot study by excluding current, recent and heavy smokers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women or men > age 18 with advanced breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Genetic Lesion detection | baseline
  To determine whether the genetic mutations in plasma DNA are reflective of the genetic mutations present in biopsies of tumor tissue obtained from ≥ 3 tumors within patients with metastatic breast cancer.

SECONDARY OUTCOMES:
Somatic genetic mutations in tumor samples | baseline
  To determine the amount of plasma DNA required to capture all somatic genetic mutations as represented in biopsied tumor samples.
Genetic heterogeneity among metastatic tumors. | baseline
  To determine the extent of genetic heterogeneity among biopsies of different metastatic tumors within patients with metastatic breast cancer.
Genetic heterogeneity between primary and metastatic breast tumors | baseline
  To determine the degree of genetic heterogeneity between primary and metastatic breast tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Chamberlin MD, Wells JD, Shee K, Bean JR, Marotti JD, Wells WA, Trask HW, Kolling FW, Bhatt A, Kaufman PA, Schwartz GN, Gemery JM, McNulty NJ, Tsapakos MJ, Barth RJ, Arrick BA, Gui J, Miller TW. Plasma DNA as a "liquid biopsy" incompletely complements tumor biopsy for identification of mutations in a case series of four patients with oligometastatic breast cancer. Breast Cancer Res Treat. 2020 Aug;182(3):665-677. doi: 10.1007/s10549-020-05714-2. Epub 2020 Jun 19. PMID 32562118